CLINICAL TRIAL: NCT04018495
Title: STimulating ImProved Health And Well-being In CysTic Fibrosis Using Integration Of Fitness Technology and Port CF.
Brief Title: STeP IT UP CF: STimulating ImProved Health And Well-being In CysTic Fibrosis
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Rose Franco, Associate Professor, Medical College of Wisconsin
Other Study IDs: 34812
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- CF patients using Fitbit for 3 months: CF patients at time of enrollment who are willing to use a fitbit tracker to measure activity and sleep during the observational period of 3 months.

SUMMARY:
STeP IT UP CF: STimulating ImProved Health And Well-being In CysTic Fibrosis Using Integration Of Fitness Technology and Port CF. A pilot in integration of wearable fitness tracker data with existing health data provided by CF foundation Patient Registry (Port CF)

DETAILED DESCRIPTION:
Cystic fibrosis patients who are willing to use an activity tracker for 3 months are invited to participate. Analysis of activity patterns and sleep patterns will be analyzed and compared to their lung function and general health as part of the routine CF center care visits during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Cystic Fibrosis
* Age >18, Cystic Fibrosis

Exclusion Criteria:

* A potential subject who meets any of the following exclusion criteria is ineligible to participate in the study.
* Those unable to commit to at least 3 months follow up for CF care from enrollment at study CF center. Inability to speak and understand English.
* Those patients without dedicated access to a smartphone, tablet, or computer with internet for syncing device and completing patient diary.
* Those patients unwilling to sign an informed consent form.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cystic fibrosis patients seen at an academic adult CF center.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose Franco, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amin R, Bean J, Burklow K, Jeffries J. The relationship between sleep disturbance and pulmonary function in stable pediatric cystic fibrosis patients. Chest. 2005 Sep;128(3):1357-63. doi: 10.1378/chest.128.3.1357. PMID 16162729
- [Background] Beattie Z, Oyang Y, Statan A, Ghoreyshi A, Pantelopoulos A, Russell A, Heneghan C. Estimation of sleep stages in a healthy adult population from optical plethysmography and accelerometer signals. Physiol Meas. 2017 Oct 31;38(11):1968-1979. doi: 10.1088/1361-6579/aa9047. PMID 29087960
- [Background] Dancey DR, Tullis ED, Heslegrave R, Thornley K, Hanly PJ. Sleep quality and daytime function in adults with cystic fibrosis and severe lung disease. Eur Respir J. 2002 Mar;19(3):504-10. doi: 10.1183/09031936.02.00088702. PMID 11936530
- [Background] de Zambotti M, Baker FC, Colrain IM. Validation of Sleep-Tracking Technology Compared with Polysomnography in Adolescents. Sleep. 2015 Sep 1;38(9):1461-8. doi: 10.5665/sleep.4990. PMID 26158896
- [Background] Gonzalez-Ortiz M, Martinez-Abundis E, Balcazar-Munoz BR, Pascoe-Gonzalez S. Effect of sleep deprivation on insulin sensitivity and cortisol concentration in healthy subjects. Diabetes Nutr Metab. 2000 Apr;13(2):80-3. PMID 10898125
- See also: Sample size requirements for estimating Pearson, Kendall and Spearman Correlations. Insufficient sleep is a public health problem. Cystic Fibrosis Trust Cystic Fibrosis Registry Report — http://www.cysticfibrosis.org.uk/the-work-we-do/uk-cf-registry/reporting-and-resources

RESULTS

PARTICIPANT FLOW:
Groups:
- CF Patients Using Fitbit for 3 Months: Fitbit tracker; is an activity tracking product that is wireless-enabled wearable technology device that measures data such as the number of steps walked, heart rate, quality of sleep, steps climbed, and other personal metrics involved in fitness
  Fitbit Tracker: Fitbit tracker; is an activity tracking product that is wireless-enabled wearable technology device that measures data such as the number of steps walked, heart rate, quality of sleep, steps climbed, and other personal metrics involved in fitness
Period: Overall Study
Arm/Group | CF Patients Using Fitbit for 3 Months
Started | 21
Completed | 20
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | CF Patients Using Fitbit for 3 Months
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Activity Tracker Utilization- Total Days of Use
Description: Descriptive statistics, such as mean for the number of days of use over the three month period
Time Frame: 3 months
Measure: Mean (Full Range); unit: Total days used
Arm/Group | CF Patients Using Fitbit for 3 Months
Number analyzed (Participants) | 21
Total days used | 85.380 [27 to 93]

2. Primary Outcome: Activity Tracker Utilization - Minutes of Sleep Per Night
Description: Descriptive statistics, such as mean for the number of minutes per sleep per night
Time Frame: 3 months
Measure: Mean (Full Range); unit: minutes of sleep per night
Arm/Group | CF Patients Using Fitbit for 3 Months
Number analyzed (Participants) | 21
minutes of sleep per night | 381.28 [0 to 983]

3. Primary Outcome: Activity Tracker Utilization - Steps Per Day
Description: Descriptive statistics, such as mean, for the number of steps per day
Time Frame: 3 months
Measure: Mean (Full Range); unit: steps/day
Arm/Group | CF Patients Using Fitbit for 3 Months
Number analyzed (Participants) | 21
steps/day | 7262.49 [0 to 30010]

4. Secondary Outcome: Integration of Cystic Fibrosis Registry Lung Function Data - Average GLI FEV1 From First to Last Day of Fitbit Wear
Description: Analyze the data trends. Forced Expiratory Volume (FEV1) reported will be used for small group analysis to compare trends with lung function mean from first to last day of wear.
Time Frame: 3 months
Measure: Mean (Full Range); unit: Percentage of Predicted FEV1
Arm/Group | CF Patients Using Fitbit for 3 Months
Number analyzed (Participants) | 21
Percentage of Predicted FEV1 | 66.535 [30.42 to 117.69]

ADVERSE EVENTS:
Time Frame: 3 months
Description: the device used is generally available to the public and is not expected to cause any adverse health events. Subjects were informed to communicate if they had any concerns related to the device.
Groups:
- Interventional - Fitbit Tracker: Fitbit tracker; is an activity tracking product that is wireless-enabled wearable technology device that measures data such as the number of steps walked, heart rate, quality of sleep, steps climbed, and other personal metrics involved in fitness
  Fitbit Tracker: Fitbit tracker; is an activity tracking product that is wireless-enabled wearable technology device that measures data such as the number of steps walked, heart rate, quality of sleep, steps climbed, and other personal metrics involved in fitness
Arm/Group | Interventional - Fitbit Tracker
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT04018495/Prot_SAP_002.pdf
  • Informed Consent Form (2020-03-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT04018495/ICF_001.pdf